CLINICAL TRIAL: NCT04092790
Title: The Identification and Prevention of Sarcopenia in Older Patients in the Acute Hospital Setting
Brief Title: Sarcopenia in Older Patients in the Acute Hospital Setting
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Principal Investigator, Tzvi Dwolatzky, Director Geriatrics, Rambam Health Care Campus
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 0053-18-RMB
Record Dates: First submitted 2019-09-15; First posted 2019-09-17 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Sarcopenia; Frailty
MeSH Terms: conditions — Sarcopenia; Frailty

STUDY DESIGN:
Intervention Model Description: Eligible subjects will be scored either as low-risk for sarcopenia-related adverse outcomes (<4) or high risk (≥4) via the SARC-F scoring system, and will be evaluated for sarcopenia of the lower limbs using a B-mode portable ultrasound machine used for standard clinical practice at the Rambam Health Care Campus. A VGD will be applied to one randomly-assigned lower limb. The VGD will be operated constantly (apart from times that the patient is being bathed or undergoing investigations or procedures) providing intermittent stimulations as outlined in the investigator brochure. On day 4, ultrasound of the lower limbs will be repeated for all subjects, with repeat imaging every subsequent second day for admissions extending beyond 4 days and a maximum of 10 days after the application of the VGD. The study will include all eligible patients in the internal department (internal medicine ward Het) who agree to participate in the study and provide written informed consent.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Virtual Gate Device (VGD) (Experimental): The Virtual Gait Device (VGD) is a technology that uses fussy-logic technology to stimulate calf muscles in synchrony with the patient's heartbeat, enabling a virtual gait in patients who have limited mobility. The stocking-like device is especially useful in older patients who are acutely hospitalized and thus at risk for sarcopenia. While physical activity and physical resistance training are well-documented as preventive measures for sarcopenia, active physical exercise is an unrealistic option for most acutely hospitalized, mobility-limited, older patients. The VGD is a practical alternative that is simple to operate. One pilot study in the orthopedics department in Hadassah Medical Center in Jerusalem, Israel was performed on patients with fractured ankles with the goal of muscle wasting prevention. The VGD will be provided by the manufacturer for use in this pilot clinical study.
  Interventions: Device: Virtual Gate Device (VGD)

INTERVENTIONS:
Device: Virtual Gate Device (VGD) — A VGD will be applied to one randomly-assigned lower limb. The VGD will be operated constantly (apart from times that the patient is being bathed or undergoing investigations or procedures) providing intermittent stimulations for a maximum of 10 days.

SUMMARY:
This study will assess whether the use of technology using the Virtual Gate Device (VGD) will prevent or minimize the development of hospital acquired Sarcopenia resulting from Immobilization.

DETAILED DESCRIPTION:
Modern advances in prevention, medical care, and treatments have resulted in an ever-increasing life expectancy and aging of the population. As a result, it is imperative that health care professionals and policy makers develop strategies and new technologies that enable older people to enjoy their advancing years in good health.

Sarcopenia, an age-related decrease in muscle mass, is a major factor in functional decline and frailty and leads to poor quality of life and increased health care costs in older age groups. Because sarcopenia is known to be exacerbated at the time of acute hospital admission, the development of new technologies for the prevention and diagnosis of sarcopenia will have important ramifications in promoting healthy aging in both the acute care and ambulatory settings.

A pilot interventional self-controlled study will be performed in an internal medicine department (internal medicine ward Het) at the Rambam Health Care Campus in Haifa.

Subjects will be evaluated for the risk of sarcopenia by acceptable screening instruments as well as B-mode portable ultrasound. They will then be treated using a stocking-like Virtual Gait Device (VGD) which will be applied to one randomly-assigned lower limb. The VGD is a technology that uses fussy-logic technology to stimulate calf muscles in synchrony with the patient's heartbeat, enabling a virtual gait in patients who have limited mobility.

Confidentiality will be achieved by applying a unique identifier to each trial subject in accordance with Good Clinical Practice standards.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients 75 years of age and older.
* Patients admitted with an acute infection (clinically from a respiratory or urinary source).
* Expected length of hospitalization of at least 4 days.
* Patients who are conscious and cognitively able to provide written informed consent as determined by a score of 0 on the 4AT scale

Exclusion Criteria:

* Male and female patients under 75 years of age.
* Expected length of hospitalization of less than 4 days.
* A condition limiting the use of the virtual gate device (VGD) due to factors relating to discomfort or safety, including but not limited to: fracture, amputation, local infection, pain, paralysis of one or both lower limbs, cardiac arrhythmia or cardiac pacemaker.
* Patients who are unable to or do not provide informed consent for participation.
* A score 1 or more on the 4AT scale.

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-04-18 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Muscle mass | Day 4 of admission or last measurement prior to discharge for a maximum of 10 days.
  Determined by B-mode ultrasound measurement.

CONTACTS AND LOCATIONS:
Overall Officials: Tzvi Dwolatzky, MD, Principal Investigator — Rambam Health Care Campus
Locations (1):
- Rambam Health Care Campus, Haifa, North, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Malmstrom TK, Miller DK, Simonsick EM, Ferrucci L, Morley JE. SARC-F: a symptom score to predict persons with sarcopenia at risk for poor functional outcomes. J Cachexia Sarcopenia Muscle. 2016 Mar;7(1):28-36. doi: 10.1002/jcsm.12048. Epub 2015 Jul 7. PMID 27066316
- [Background] Ticinesi A, Meschi T, Narici MV, Lauretani F, Maggio M. Muscle Ultrasound and Sarcopenia in Older Individuals: A Clinical Perspective. J Am Med Dir Assoc. 2017 Apr 1;18(4):290-300. doi: 10.1016/j.jamda.2016.11.013. Epub 2017 Feb 13. PMID 28202349
- [Background] Maddocks M, Nolan CM, Man WD, Polkey MI, Hart N, Gao W, Rafferty GF, Moxham J, Higginson IJ. Neuromuscular electrical stimulation to improve exercise capacity in patients with severe COPD: a randomised double-blind, placebo-controlled trial. Lancet Respir Med. 2016 Jan;4(1):27-36. doi: 10.1016/S2213-2600(15)00503-2. Epub 2015 Dec 15. PMID 26701362
- See also: 4AT- Rapid clinical test for delirium — https://www.the4at.com